CLINICAL TRIAL: NCT07014137
Title: A Phase II Trial of ABSK043, an Oral PD-L1 Inhibitor, in Patients With Angiogenic Sarcomas
Brief Title: A Trial of ABSK043, an Oral PD-L1 Inhibitor, in Patients With Angiogenic Sarcomas
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SARC-005
Record Dates: First submitted 2025-05-01; First posted 2025-06-10 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- open label - Anti-PD-L1 (ABSK043) (Other)
  Interventions: Drug: ABSK043 single agent

INTERVENTIONS:
Drug: ABSK043 single agent — ABSK043 BID continuously for 28 day cycle
  Other Names: ABSK043

SUMMARY:
ABSK043 is a new type of experimental drug that blocks a protein called programmed cell death ligand 1 (PD-L1), which is important in controlling the body's response to harmful substances including cancer cells. By blocking PD-L1 from working, ABSK043 may allow the body's immune system to recognize and kill cancer cells.

ABSK043 is considered "experimental" because it has not been approved for sale by Health Canada. Health Canada has approved the study drug to be administered in this research study.

The main purposes of this study are:

* To see if patients with your type of cancer benefit from ABSK043.
* To evaluate the safety and tolerability of ABSK043.
* To identify biomarkers (Biological flags used to measure disease progress or drug effect.) in tumor tissues or blood that might help identify patients whose cancers respond to ABSK043, and which patients may develop side effects from these study drugs. Examples of biomarkers include the type of white blood cells in your tumor or proteins in your blood.

It is anticipated that about 20 people will take part in this study from the Princess Margaret Cancer Centre.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Be >18 years of age on day of signing informed consent.
3. Have one of the following advanced (unresectable and/or metastatic) solid tumor indications:

   1. Intimal sarcoma
   2. Head and neck angiosarcoma
   3. Epithelioid hemangioendothelioma (EHE)
4. Have measurable disease based on RECIST v1.1.
5. Have a performance status of 0, 1, or 2 on the ECOG Performance Scale.
6. Have the ability to swallow and retain orally administered medications.
7. Demonstrate adequate organ function as defined in Table 1, all screening labs should be performed within 10 days of treatment initiation.
8. Female subject of childbearing potential should have a negative serum pregnancy within 72 hours prior to receiving the first dose of study medication.
9. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (Reference Section 7.1.4.3). Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
10. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

The subject must be excluded from participating in the trial if the subject:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. Use of steroids at physiological dose is allowed (i.e. less than or equal to prednisone 10mg per day)
3. Has had prior treatment with any anti-PD-1, anti-PD-L1 or other antibodies specifically targeting the immune checkpoint pathways.
4. Has had a prior anti-cancer monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
5. Has active gastrointestinal condition that may affect the absorption of ABSK043, according to investigator.
6. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy or alopecia are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
7. Has a known additional malignancy within the last 3 years or continues to receive antineoplastic treatment after curative intent surgery. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
8. Has known active central nervous system (CNS) metastases and/or leptomeningeal disease. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include leptomeningeal disease which is excluded regardless of clinical stability.
9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
10. Has known history of, or any evidence of active, non-infectious pneumonitis.
11. Has evidence of interstitial lung disease.
12. Has an active infection requiring systemic treatment.
13. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
14. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
15. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
16. Has a known history of Human Immunodeficiency Virus (HIV) with detectable viral load.
17. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
18. A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 milliseconds (ms)).
19. A history of additional risk factors for torsades de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).
20. The use of concomitant medications that prolong the QT/QTc interval.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2026-03-02 (Estimated); Study Completion 2026-03-02 (Estimated)

PRIMARY OUTCOMES:
overall response rate of ABSK043 therapy in angiogenic sarcomas (i.e. intimal, head/neck angiosarcoma, and EHE) | through study completion, an average of 1 year
  To determine the overall response rate of ABSK043 therapy in angiogenic sarcomas (i.e. intimal, head/neck angiosarcoma, and EHE). Tumor response as defined by the investigator-assessed Response Evaluation Criteria in Solid Tumors criteria version 1.1 (RECIST v 1.1) for solid tumor histology.

CONTACTS AND LOCATIONS:
Locations (1):
- UHN- Princess Margaret Cancer Center, Toronto, Ontario, Canada